CLINICAL TRIAL: NCT03468283
Title: A Randomized, Controlled, Open-label Study to Evaluate the Efficacy of Smartphone Application in Patients With Type 2 Diabetes
Brief Title: Smartphone Application for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Cheol-Young Park, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KBC12093
Record Dates: First submitted 2018-03-01; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Mobile healthcare; Health Services Research; Community Health Services; Diabetes self-management education
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention was the addition of mobile healthcare-based diabetes self-management education, which consisted of "mobile application for diabetes" and individualized regular message feedback sent by healthcare professionals, to current diabetes management.
  Interventions: Other: mobile application for diabetes
- control (No Intervention): Participants of control group maintained previous diabetes management in Kangbuk Samsung Hospital throughout this study. Providers were not involved with patient prescriptions.

INTERVENTIONS:
Other: mobile application for diabetes — Intervention was mobile application and individualized regular message feedback sent by healthcare professionals.
  Arms: Intervention

SUMMARY:
Since diabetes is a chronic disease closely related to unhealthy lifestyle, the improvement and management of living habits are as significant as medical care with regard to the disease. In addition, this is regarded as the most effective method for prevention and treatment of diabetes. However, many diabetic patients are now reported to lack proper management in Korea with a low level of compliance with treatment instruction. In that sense, it is urgently necessary to develop a program in which diabetic patients are able to effectively manage their own blood glucose at home, and to grasp the real state of self-blood glucose measurement. Accordingly, a system to manage diabetes using electronic equipment such as mobile phone or the Internet is currently being developed and studied, for the effective management of diabetes with the help of highly evolving information technology. These investigators have developed a diabetes management program that provides an optimal solution based on a mobile device and software, so that individual patients can undergo a regular blood glucose test and achieve improvement and constant management of living habits by being properly informed of how to manage diabetes. This clinical study was designed to evaluate the effectiveness and efficacy of the application through the comparison between usual medical care and additional care using the smartphone application, targeting patients with type 2 diabetes who lack blood glucose control. This study is targeted at the subjects who are being treated at this hospital's endocrinology, are using a smartphone, and voluntarily signed the informed consent form (ICF). The subjects who pass the subject eligibility evaluation provide information regarding assessment items and demographic information using the smartphone application and questionnaire. Based on the information given by subjects, the medical team offers a management system that supports and improves the existing treatment process of diabetes using the application developed on its own. The feasibility and effectiveness of the management using the application are evaluated through the result values of the laboratory tests performed during the subject's usual medical care.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 19 years;
* android smartphone users;
* no changes in medication for diabetes for at least 6 months;
* HbA1c levels ≥6.5% within the last 3 months.

Exclusion Criteria:

* currently had serious concomitant disease other than diabetes (n=1); malignancy-related histories on admission, myocardial infarction, cerebral infarction or organ transplantation;
* pregnant or had plans for pregnancy within 6 months;
* plans to participate in other clinical studies or illiteracy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-08-07 (Actual); Primary Completion 2013-02-06 (Actual); Study Completion 2013-03-13 (Actual)

PRIMARY OUTCOMES:
hemoglobin A1c levels | at six months
  serum glycated hemoglobin levels

SECONDARY OUTCOMES:
body mass index | at six months
  The changes in body mass index
blood pressure | at six months
  The changes in blood pressure
serum triglyceride | at six months
  The changes in serum triglyceride levels
serum high-density lipoprotein cholesterol | at six months
  The changes in serum high-density lipoprotein cholesterol levels
serum low-density lipoprotein cholesterol | at six months
  The changes in serum low-density lipoprotein cholesterol levels
Summary of Diabetes Self-Care Activities Questionnaire | at six months
  scores of Summary of Diabetes Self-Care Activities Questionnaire to measure the current status of diabetic patients' self-care activities (diet, exercise, blood glucose, foot care, and smoking) with each scale of 0 to 7 points.
Audit of Diabetes Dependent Quality of Life | at six months
  scores of Audit of Diabetes Dependent Quality of Life to measure effects of diabetes on the quality of patients' life with each scale of -9 to +3 points.
the Korean version of the Appraisal of Diabetes Scale | at six months
  scores of the Korean version of the Appraisal of Diabetes Scale to measure how diabetic patients recognize about the disease with each scale of 1 to 5 points.
the Problem Areas in Diabetes | at six months
  scores of the Problem Areas in Diabetes to measure level of stress related to diabetes with each scale of 0 to 4 points.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee DY, Yoo SH, Min KP, Park CY. Effect of Voluntary Participation on Mobile Health Care in Diabetes Management: Randomized Controlled Open-Label Trial. JMIR Mhealth Uhealth. 2020 Sep 18;8(9):e19153. doi: 10.2196/19153. PMID 32945775